CLINICAL TRIAL: NCT06392880
Title: Comparison of the Effects of Floss Taping and Mulligan Mobilization on Ankle Joint Movement, Vertical Jump, Gait and Balance in Healthy Young Adults
Brief Title: Comparison of Floss Band Application and Mulligan Mobilization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Associate Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2024/02
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Health, Subjective
Keywords: ankle motion; gait; vertical jump; balance

STUDY DESIGN:
Intervention Model Description: This study features a balanced cross-over design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Floss Band (Experimental): A floss band will be applied to the ankle joint and the participant will practice various weight-bearing active ankle motions simultaneously.
  Interventions: Other: Floss Band; Other: Mulligan Mobilization; Other: Control
- Mulligan mobilization (Experimental): Mulligan mobilization will be applied to the ankle joint and the participant will practice various weight-bearing active ankle motions simultaneously.
  Interventions: Other: Floss Band; Other: Mulligan Mobilization; Other: Control
- Control (Other): Participants will practice various weight-bearing active ankle motions.
  Interventions: Other: Floss Band; Other: Mulligan Mobilization; Other: Control

INTERVENTIONS:
Other: Floss Band — A floss band will be applied to the ankle joint and the participant will practice various weight-bearing active ankle motions simultaneously.
Other: Mulligan Mobilization — Mulligan mobilization will be applied to the ankle joint and the participant will practice various weight-bearing active ankle motions simultaneously.
Other: Control — Participants will practice various weight-bearing active ankle motions simultaneously.

SUMMARY:
This study will investigate the effects of Floss band application and Mulligan mobilization on ankle range of motion, vertical jump, gait and balance in active healthy young adults.

DETAILED DESCRIPTION:
The effects of floss band application and mulligan mobilization on ankle range of motion, vertical jump, gait, and balance in active healthy young adults are unclear or limited due to a lack of studies. There are also no other studies comparing the two interventions in healthy young adults. Therefore, this study will investigate the effects of Floss band application and Mulligan mobilization on ankle range of motion, vertical jump, gait, and balance in active healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-24 years,
* Not having any known disease
* Being recreationally active
* Body mass index between 18.5 and 29.9 kg/m2

Exclusion Criteria:

* Presence of cardiovascular, rheumatic, dermatologic, orthopedic or neurologic diseases
* History of injury or trauma in the last 6 months

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-05-14 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
Passive ankle joint range of motion | The assessment will be conducted before and immediately after the interventions.
  Passive ankle range of motion will be evaluated by taking photographs. Measurements will be made with Image-J program on the photograph.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, PhD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Derived] Horata E, Tasvuran Horata E, Kanyilmaz AN, Solak HI. Comparison of tissue flossing and mobilization with movement effects on motion, vertical jump, gait, and balance. BMC Sports Sci Med Rehabil. 2026 Jan 19. doi: 10.1186/s13102-026-01533-y. Online ahead of print. PMID 41555334